CLINICAL TRIAL: NCT01380223
Title: A First-in-Man, Phase I, Double-Blind, Randomized, Four-Way Crossover, Placebo-Controlled, Dose-Escalation, Pharmacokinetic and Pharmacodynamic Study of CK-1827452 (Omecamtiv Mecarbil) in Healthy Volunteers
Brief Title: A Pharmacokinetic and Pharmacodynamic Study of Omecamtiv Mecarbil in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CY 1111; 2005-001886-32 (EudraCT Number)
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — omecamtiv mecarbil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose-escalation Cohort 1 (Experimental): 4 treatment periods consisting of a 2 hour placebo infusion (single blind) followed by a 6 hour infusion of study drug or placebo. Each subject will receive 3 active ascending doses of study drug and 1 dose of placebo randomized into the sequence of escalating doses in a double-blind manner. Treatment periods occur at least 7 days apart.
  Interventions: Drug: placebo; Drug: omecamtiv mecarbil
- Dose-escalation Cohort 2 (Experimental): 4 treatment periods consisting of a 2 hour placebo infusion (single blind) followed by a 6 hour infusion of study drug or placebo. Each subject will receive 3 active ascending doses of study drug and 1 dose of placebo randomized into the sequence of escalating doses in a double-blind manner. Treatment periods occur at least 7 days apart.
  Interventions: Drug: placebo; Drug: omecamtiv mecarbil
- Dose-escalation Cohort 3 (Experimental): 4 treatment periods consisting of a 2 hour placebo infusion (single blind) followed by a 6 hour infusion of study drug or placebo. Each subject will receive 3 active ascending doses of study drug and 1 dose of placebo randomized into the sequence of escalating doses in a double-blind manner. Treatment periods occur at least 7 days apart.
  Interventions: Drug: placebo; Drug: omecamtiv mecarbil
- Dose-escalation Cohort 4 (Experimental): 4 treatment periods consisting of a 2 hour placebo infusion (single blind) followed by a 6 hour infusion of study drug or placebo. Each subject will receive 3 active ascending doses of study drug and 1 dose of placebo randomized into the sequence of escalating doses in a double-blind manner. Treatment periods occur at least 7 days apart.
  Interventions: Drug: placebo; Drug: omecamtiv mecarbil

INTERVENTIONS:
Drug: placebo — I.V. infusion of placebo for 8 hr
Drug: omecamtiv mecarbil — I.V. infusion of placebo for 2 hr followed by 6 hr infusion of omecamtiv mecarbil at 0.005 mg/kg/hr
  Other Names: CK-1827452, AMG 423
  Arms: Dose-escalation Cohort 1
Drug: omecamtiv mecarbil — I.V. infusion of placebo for 2 hr followed by 6 hr infusion of omecamtiv mecarbil at 0.015 mg/kg/hr
  Other Names: CK-1827452, AMG 423
  Arms: Dose-escalation Cohort 1
Drug: omecamtiv mecarbil — I.V. infusion of placebo for 2 hr followed by 6 hr infusion of omecamtiv mecarbil at 0.025 mg/kg/hr
  Other Names: CK-1827452, AMG 423
  Arms: Dose-escalation Cohort 1; Dose-escalation Cohort 2
Drug: omecamtiv mecarbil — I.V. infusion of placebo for 2 hr followed by 6 hr infusion of omecamtiv mecarbil at 0.0625 mg/kg/hr
  Other Names: CK-1827452, AMG 423
  Arms: Dose-escalation Cohort 2
Drug: omecamtiv mecarbil — I.V. infusion of placebo for 2 hr followed by 6 hr infusion of omecamtiv mecarbil at 0.125 mg/kg/hr
  Other Names: CK-1827452, AMG 423
  Arms: Dose-escalation Cohort 2; Dose-escalation Cohort 3
Drug: omecamtiv mecarbil — I.V. infusion of placebo for 2 hr followed by 6 hr infusion of omecamtiv mecarbil at 0.25 mg/kg/hr
  Other Names: CK-1827452, AMG 423
  Arms: Dose-escalation Cohort 3
Drug: omecamtiv mecarbil — I.V. infusion of placebo for 2 hr followed by 6 hr infusion of omecamtiv mecarbil at 0.5 mg/kg/hr
  Other Names: CK-1827452, AMG 423
  Arms: Dose-escalation Cohort 3; Dose-escalation Cohort 4
Drug: omecamtiv mecarbil — I.V. infusion of placebo for 2 hr followed by 6 hr infusion of omecamtiv mecarbil at 1.0 mg/kg/hr
  Other Names: CK-1827452, AMG 423
  Arms: Dose-escalation Cohort 4
Drug: omecamtiv mecarbil — I.V. infusion of placebo for 2 hr followed by 6 hr infusion of omecamtiv mecarbil at 0.75 mg/kg/hr (dose reduced)
  Other Names: CK-1827452, AMG 423
  Arms: Dose-escalation Cohort 4
Drug: omecamtiv mecarbil — I.V. infusion of placebo for 2 hr followed by 6 hr infusion of omecamtiv mecarbil at 0.625 mg/kg/hr (dose reduced)
  Other Names: CK-1827452, AMG 423
  Arms: Dose-escalation Cohort 4

SUMMARY:
This study will assess the safety, tolerability, and pharmacodynamics of omecamtiv mecarbil infusion in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male
2. Subject is aged between 18 and 50 years inclusive.
3. Subject has given signed informed consent.
4. Subject's Body Mass Index (BMI) is between 18 and 30 kg/m2 inclusive.
5. Subject weighs less than 100 kg.
6. Subject is considered to be in good health in the opinion of the investigator, as determined by:

   1. A pre-study physical examination with no clinically significant abnormalities.
   2. Vital signs within normal ranges (supine after 3 minutes rest - heart rate: 40 to 80 bpm; systolic BP: 100 to 140 mmHg; diastolic BP: 50-90 mmHg; respiration rate: 8 to 18 breaths per minute; oxygen saturation: 96-100%)
   3. An ECG with no clinically significant abnormalities.
7. Subject's pre-study clinical laboratory findings are within normal range or if outside of the normal range not deemed clinically significant in the opinion of the investigator.
8. Cardiac troponin I is less than the upper limit of the laboratory reference range.
9. A screening echocardiogram demonstrates normal cardiac function, an ejection fraction of between 40% and 70% with no significant valvular regurgitation (grade 1) and/or stenosis and images are deemed to be of good quality by the sonographer.

Exclusion Criteria:

1. Subject has had a clinically significant illness in the four weeks before screening.
2. Use of prescribed mediations in the 3 weeks prior to dosing or over-the-counter preparations (including vitamin supplements and herbal remedies) for 7 days prior to dosing, except paracetamol which will be allowed up to 48 hours prior to dosing.
3. Subject has a significant history of drug/solvent abuse or a positive drugs of abuse test at screening.
4. Subject with a history of alcohol abuse or currently drinks in excess of 28 units per week.
5. Subject smokes more than 5 cigarettes (or equivalent) per day.
6. Subject is not willing to refrain from caffeine/xanthine containing products from 48 hours prior to the screening medical and admission on Day -1 until the post study medical.
7. Subject is in the opinion of the investigator not suitable to participate in the study.
8. Subject who has participated in any clinical study with an investigational drug/device within three months prior to the first day of dosing.
9. Subject who has a positive result of HIV screen, Hepatitis B screen or Hepatitis C screen.
10. Subject has had a serious adverse reaction or significant hypersensitivity to any drug.
11. Subject has donated 500 ml or more of blood within the month prior to screening.
12. Subject has a history of cardiovascular disease or family history of premature cardiovascular disease or death.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2005-08; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Omecamtiv Mecarbil in Healthy Volunteers | 2 days
  The highest infusion rate tolerated by at least eight subjects. A dose was intolerable if: 1) the pattern of intolerance clearly distinguished active drug from placebo, or 2) the number of subjects intolerant of the dose level in question was at least 3 more than the number of subjects intolerant of placebo.

SECONDARY OUTCOMES:
Change From Baseline of Systolic Ejection Time at Various Omecamtiv Mecarbil Infusion Rates | 1 day
  Pooled analysis of the echocardiographic measure systolic ejection time. The systolic ejection time is the period during which the aortic valve is open and blood is flowing across the valve. Echocardiograms from cohorts 1,2,3,4 were binned into either placebo group or groups based on infusion rate of omecamtiv mecarbil.
Change From Baseline of Fractional Shortening at Various Omecamtiv Mecarbil Infusion Rates | 1 day
  Pooled analysis of the echocardiographic measure fractional shortening. Fractional shortening is the percentage of change from baseline in the left ventricular cavity dimension with systole. Echocardiograms from cohorts 1,2,3,4 were binned into either placebo group or groups based on infusion rate of omecamtiv mecarbil.

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Development Solutions, Manchester, England, United Kingdom

REFERENCES:
- [Derived] Vu T, Ma P, Xiao JJ, Wang YM, Malik FI, Chow AT. Population pharmacokinetic-pharmacodynamic modeling of omecamtiv mecarbil, a cardiac myosin activator, in healthy volunteers and patients with stable heart failure. J Clin Pharmacol. 2015 Nov;55(11):1236-47. doi: 10.1002/jcph.538. Epub 2015 Jul 14. PMID 25951506
- [Derived] Teerlink JR, Clarke CP, Saikali KG, Lee JH, Chen MM, Escandon RD, Elliott L, Bee R, Habibzadeh MR, Goldman JH, Schiller NB, Malik FI, Wolff AA. Dose-dependent augmentation of cardiac systolic function with the selective cardiac myosin activator, omecamtiv mecarbil: a first-in-man study. Lancet. 2011 Aug 20;378(9792):667-75. doi: 10.1016/S0140-6736(11)61219-1. PMID 21856480